CLINICAL TRIAL: NCT02670694
Title: Sleep Abnormalities in Rare Genetic Disorders: Angelman Syndrome, Rett Syndrome, and Prader Willi
Brief Title: Sleep Abnormalities in Rare Genetic Disorders: AS, RTT, and PW
Acronym: RDCRN
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: Boston Children's Hospital (Other); University of California, San Diego (Other); Greenwood Genetic Center (Other); University of Florida (Other); Vanderbilt University (Other); University of Kansas Medical Center (Other); University of California, Irvine (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Daniel Glaze, Principal Investigator, Baylor College of Medicine
Other Study IDs: H-26535
Record Dates: First submitted 2015-11-06; First posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Rett Syndrome; Prader-Willi Syndrome; Angelman Syndrome; Sleep Problems
Keywords: Rett Syndrome; Prader-Willi Syndrome; Angelman Syndrome; Sleep Problems
MeSH Terms: conditions — Rett Syndrome; Prader-Willi Syndrome; Angelman Syndrome; Parasomnias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Rett Syndrome: Children and adolescents, age between 0-19 years, with clinical diagnosis of Rett Syndrome; currently enrolled in the Rare Disease Clinical Research Network registry.
- Angelman's Syndrome: Children and adolescents, age between 0-19 years, with clinical diagnosis of Angelman's Syndrome; currently enrolled in the Rare Disease Clinical Research Network registry.
- Prader-Willi Syndrome: Children and adolescents, age between 0-19 years, with clinical diagnosis of Prader-Willi Syndrome; currently enrolled in the Rare Disease Clinical Research Network registry.
- Control: Siblings of RTT, AS and PW subjects will serve as control subjects.

SUMMARY:
This study will investigate sleep behavior in subjects with Angelman Syndrome, Rett Syndrome or Prader-Willi Syndrome.

The study will also investigate sleep behavior in healthy siblings of subjects with Angelman Syndrome, Rett Syndrome or Prader-Willi Syndrome. These individuals will serve as control subjects.

The study will use questionnaires designed to identify sleep disorders and how they affect behavior and quality of life.

The principal goals of this study are:

1. To see how common sleep disorders are in individuals with Angelman Syndrome, Rett Syndrome or Prader-Willi Syndrome;
2. To see how sleep disorders affect behavior in these individuals;
3. To see whether sleep disorders and related behavior problems improve or worsen with age;
4. To see how specific disease conditions relate to sleep disorders and how bad the sleep disorders are;
5. To develop new treatment options to improve quality of life and behavior issues; and
6. To evaluate current treatment options to improve sleep problems in these individuals.

DETAILED DESCRIPTION:
Subjects with AS, RTT or PWS and normal siblings (controls) will be recruited for study participation.

Subjects will be recruited from the Rare Disease Clinical Research Network (RDCRN) consortium registries for AS, RTT and PWS. The RDCRN registries provide listings of individuals currently enrolled in the RDCRN along with clinical and genetic diagnosis, medical history and contact information.

The RDCRN consortium sites for AS, RTT and PWS will participate in the study. These sites will recruit study participants, obtain informed consent and administer the sleep questionnaires. Institutional Review Board (IRB) approval will be obtained at each RDCRN consortium site.

"Subjects" is defined as those children with a diagnosis of AS, PWS, and RTT. Subjects will be divided into separate study arms based upon their medical diagnosis. Study arms will consist of: 1) AS group, 2) PWS group, 3) RTT group, and 4) control group. "Control group" is defined as normal healthy siblings of subjects.

Study participants and parents/guardians will be asked to complete the study questionnaires during the clinic visit. The questionnaires are brief and should not be difficult to complete. It is anticipated that the questionnaires can be completed in 15-30 minutes. If parents are unable to complete the questionnaires at the time of their scheduled clinic visit they will be asked to take the questionnaires home to complete and to mail them back to the research team. When the research team receives the returned questionnaires they will be reviewed for completion. If questions are skipped or left blank, a member of the research team will call the family to complete the missed questions over the phone.

Parents/guardians are allowed to answer the questions on behalf of the study participants and will be asked to answer all the questions for each age-appropriate questionnaire in order for the responses to be scored correctly. Subjects with AS, RTT and PWS and normal siblings will complete the same questionnaire forms.

Study participants will be administered the questionnaires again in 12-24 months at a follow-up RDCRN clinic visit or by mail to assess the natural history of their sleep behavior and any sleep disorders.

Study participants identified as having a potential severe sleep disorder based on questionnaire responses will be contacted or sent a letter by the study investigators and advised to see a sleep specialist for further evaluation.

Potential "Subjects" must be members of the RDCRN consortium registries with available contact and clinical diagnostic information on file. These individuals will be invited to participate in the study at their next regularly scheduled RDCRN visit.

Study recruitment will continue for one year. Subjects with a clinical diagnosis of AS, RTT or PWS, or normal siblings of these individuals will be recruited for study participation.

The sample size of study participants, including controls, will be based upon the number of individuals currently enrolled in the RDCRN consortium registries. Currently the combined number of individuals in the AS, RTT and PWS RDCRN consortium registries is 1082. The breakdown by disorder is: 678 RTT, 172 AS, 141 PWS. Final sample size will be the total number of subjects consented during the one year recruitment period. A projected enrollment total would be approximately 1,000 total individuals ( 500 subjects including 300 RTT, 100 AS, 100 PWS & 500 controls).

ELIGIBILITY:
Inclusion Criteria:

Eligible Inclusion Criteria - Subjects

1. Enrollment in a RDCRN consortium registry for either AS, RTT or PWS.
2. Have a clinical diagnosis of AS, RTT or PWS, or be a normal sibling of an individual with AS, RTT or PWS who is enrolled in the study.
3. Be between 0 to18 years of age inclusive.
4. Be English-speaking (study questionnaires will only be available in English).

Inclusion Criteria - Controls

1. Must have a sibling with either AS, RTT or PWS enrolled in the study.
2. Must not have a diagnosis of any neurological disorder.
3. Be between 0 to18 years of age inclusive
4. Be English-speaking (study questionnaires will only be available in English).

Exclusion Criteria:

Exclusion Criteria - Subjects

1. No clinical diagnosis of AS, RTT, or PWS.
2. Diagnosis of a severe genetic disorder in addition to AS, RTT, or PWS.
3. Be over 18 years of age inclusive.

Exclusion Criteria - Controls

1. Diagnosis of a neurological disorder.
2. Diagnosis of a severe genetic disorder.
3. Be over 19 years of age inclusive.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This research study will investigate sleep behavior in the rare neurological disorders Angelman Syndrome (AS), Rett Syndrome (RTT) and Prader-Willi Syndrome (PWS).
Sampling Method: Non-Probability Sample
Enrollment: 804 (Actual)
Dates: Start 2011-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in sleep behavior as measured by the child's sleep habits questionnaire (CSHQ) for Rett Syndrome, Angleman and control group | Change from Baseline sleep behaviors at 24 months

SECONDARY OUTCOMES:
Pediatric Sleep Questionnaire (PSQ) - Sleep Disordered Breathing Subscale | Change from Baseline sleep behaviors at 24 months
Child's Sleep Habits Questionnaire (CSHQ) (ages 0-19) | Change from Baseline sleep behaviors at 24 months
Pediatric Daytime Sleepiness Scale (PDSS) (ages 6-19) | Change from Baseline sleep behaviors at 24 months
Cleveland Adolescent Sleepiness Questionnaire (CASQ) (ages 6-19) | Change from Baseline sleep behaviors at 24 months
Narcolepsy Questionnaire (ages 0-19) | Change from Baseline sleep behaviors at 24 months
Unique Questionnaire (ages 0-19) | Change from Baseline sleep behaviors at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Glaze, MD, Study Chair — Baylor College of Medicine; Alan Percy, MD, Study Director — University of Alabama at Birmingham; Sanjeev Kothare, MD, Principal Investigator — Harvard Medical School, Children's Hospital Boston
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, Irvine Medical Center, Irvine, California
  - Rady Children's Hospital, San Diego, California
  - University of Florida College of Medicine, Gainesville, Florida
  - Kansas University Medical Center, Kansas City, Kansas
  - Children's Hospital Boston, Boston, Massachusetts
  - Greenwood Genetic Center, Greenwood, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No